CLINICAL TRIAL: NCT03607435
Title: A Clinical Study to Collect Calibration & Performance Data of the KBS Systems 1.0 Non-Invasive Glucose Monitoring Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Florida Hospital Tampa Bay Division (Other)
Collaborators: Kaligia Biosciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KBS002
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test Article Scanning (Experimental): Spectroscopy for Analyte Quantification
  Interventions: Device: Spectroscopy for Analyte Quantification

INTERVENTIONS:
Device: Spectroscopy for Analyte Quantification — Diabetic hospital staff participants subjected to the KBS-1 device (Test Article #01) will have a finger on their left hand pricked with a lancet and their blood glucose level read by a POC glucose monitor (Control Article #02). Next, they will have their interstitial fluid glucose level spectroscopically scanned from the palm of their left hand using the KBS-1 device, and blood (approximately 40µl), collected from their finger prick site, will be spectroscopically scanned using the RBA-1 device (Test Article #02). Hospital patients subjected to the RBA-1 device, who must already be prescribed a hospital lab blood test by their physician, will have approximately 40µl of their blood, collected from the venipuncture site, spectroscopically scanned using the RBA-1 device (Test Article #02).

SUMMARY:
The purpose of this study is to calibrate the performance of the KBS-1 non-invasive glucose monitoring device with diabetic people when compared to that of the standard method currently used in the clinical setting for prescription point-of-care (POC) blood glucose monitoring. The secondary purpose of this study is to calibrate the performance of the RBA-1 minimally invasive bodily fluid analyte analyzer device when compared to the results from a prescription POC blood glucose monitoring device and/or standard hospital laboratory blood test.

The objective of this study is to collect non-invasive in vivo, and potentially in vitro, spectral measurements of interstitial fluid glucose from underneath the skin of the palm of the hand (Test Article #01), and potentially the blood, respectively, from diabetic adult hospital staff participants, and to collect in vitro spectral measurements of venous blood tested from adult hospital patients with or without diabetes (Test Article #02) and compare them to POC blood glucose monitor values and analyte measurements conducted by a hospital laboratory (Control Article #01 procedure), respectively.

The comparison of the results obtained from the different analytical methods will be used to calibrate and refine the glucose, and other, analyte level calculation algorithms of the Test Article systems.

ELIGIBILITY:
Inclusion Criteria:

Ideally, all enrolled participants will represent an ethnically diverse population with as close to an even ratio of males to females as possible.

1) Age ≥ 21 years. 2) Willingness and ability to provide informed consent.

* Additional inclusion criteria specific to KBS-1 (Test Article #01) testing:

  1) Diabetic hospital staff
* Additional inclusion criteria specific to RBA-1 (Test Article #02) testing:

  1. Hospital patients with a physician prescribed hospital laboratory blood test.
  2. Diabetic hospital staff

     Exclusion Criteria:

     The following exclusion criteria apply to all prospective study participants.

  <!-- -->

  1. A member of a vulnerable population (i.e. children, pregnant women, prisoners, etc.)
  2. People with clotting factor disorders and/or currently taking anticoagulation medication.
  3. Has any other medical condition that, in the opinion of the Investigator, would interfere with the person's participation in this study (i.e. double arm amputee).
* Additional exclusion criteria specific to KBS-1 (Test Article #01) testing:

  1. Any skin abnormalities or tattoos located on the palm(s) of the hand(s). The left palm is preferred for this study; however, the right palm can be used if the left palm is excluded.
  2. Parkinson's disease, dyskinesia, tremors, or similar that may make it challenging for said person to hold their hand on the device in a still and stable manner.
* Additional inclusion criteria specific to RBA-1 (Test Article #02) testing:

  1. Patient is in isolation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Calibration of the KBS-1 Test Article using the POC Control data for comparison. | The test article and control article procedure together will take approximately 10 - 15 minutes of the research participant's time.
  The data gathered by the Test Article procedures will be compared to the data gathered by the POC Control Article procedure in order to accomplish:
  * Comparative analysis of the Test data against the Control data.
  * Test Article calibration and aid in Test Article machine learning. This is being requested to achieve calibration of the test articles, and aid in test article machine learning for glucose level calculations.

SECONDARY OUTCOMES:
Research Subject Assessment | The assessment will take place immediately at the conclusion of the KBS-1 and POC glucose monitoring procedure and will take approximately 1 minute of the research participant's time.
  The research subjects will be questioned on the presence (Y or N) of any pain or discomfort related to the KBS-1 test article procedure, as well as ease of use and acceptability (1-5 rating scale, 1=bad, 5=excellent).
Calibration of the RBA-1 Test Article using the hospital lab test Control data and POC blood glucose monitor Control data for comparison. | The test and control article procedure together will take approximately 10 minutes of a research participant's time.
  The data gathered by the Test Article procedure will be compared to the data gathered by the Control Article procedure(s) in order to accomplish:
  * Comparative analysis of the Test data against the Control data.
  * Test Article calibration and aid in Test Article machine learning. The analyte data from the hospital lab is being requested to achieve calibration of the test article, and aid in test article machine learning, for these analytes.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Stocker, PhD, Principal Investigator — Kaligia Biosciences, LLC
Locations (1):
- Florida Hospital Tampa, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: American Diabetes Association — http://www.diabetes.org/diabetes-basics/statistics/?loc=db-slabnav